CLINICAL TRIAL: NCT07324265
Title: A Cluster-Randomized Pilot Trial of a School-Based Mental Health Literacy Program With and Without an Indirect Contact Component for 5th-Grade Students
Brief Title: Pilot Cluster RCT of an Indirect Contact Mental Health Literacy Program for 5th-Grade Students
Acronym: SMHLP-IC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo University (Other)
Responsible Party: Principal Investigator, Nobuko Demura, PhD Student, Graduate School of Education, Tokyo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SMHLP-IC-2025
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Mental Health Literacy; Stigma (Social Distance); Help-seeking Intention
Keywords: Mental health literacy; Stigma reduction; Indirect contact; Social distance; Help-seeking intentions; School-based intervention; Elementary school students
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Intervention Model Description: Cluster-randomized parallel-group design with four 5th-grade classes assigned (2:2) to intervention or control conditions. Randomization occurs at the class level within the same school.
Who Masked: Participant
Masking Description: Students were not informed whether they were in the intervention or control class. Classroom teachers delivering the lesson were aware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indirect Contact (Experimental): A 45-minute school-based mental health literacy lesson that includes an animated video, educational slides, and an additional indirect contact component. The indirect contact consists of a teacher-delivered story about a well-known soccer player who experienced and recovered from a mental health condition.
  Interventions: Behavioral: Indirect Contact
- Standard MHL Lesson Only (Active Comparator): A 45-minute standard mental health literacy lesson that includes an animated educational video and slides. This lesson does not include the indirect contact story component.
  Interventions: Behavioral: Standard MHL Lesson Only

INTERVENTIONS:
Behavioral: Indirect Contact — A 45-minute school-based mental health literacy lesson including an animated video, educational slides, and an additional indirect contact component in the form of a teacher-delivered story about a well-known soccer player who experienced and recovered from a mental health condition.
  Arms: Indirect Contact
Behavioral: Standard MHL Lesson Only — A 45-minute standard mental health literacy lesson including an animated educational video and slides, without the indirect contact story component.
  Arms: Standard MHL Lesson Only

SUMMARY:
This cluster-randomized pilot trial will evaluate the preliminary effects and feasibility of adding an indirect contact component to a school-based mental health literacy (MHL) lesson for 5th-grade students in a public elementary school in Tokyo, Japan. Four 5th-grade classes (approximately 150 students in total) will be randomized by class (two classes per arm). All students will receive a 45-minute lesson that includes an animated video and educational slides. In the intervention arm, teachers will additionally introduce a short story about a well-known soccer player who experienced and recovered from a mental health condition, serving as an indirect contact element. The control arm will receive the standard lesson without this component.

Students will complete questionnaires at baseline (T1), immediately after the lesson (T2), and 2-3 months later (T3). The primary outcome is vignette-based social distance toward a peer with mental health problems. Secondary outcomes include mental health knowledge, help-seeking intentions, perceived need for help, intended sources of help. As a pilot study with only four clusters, the trial is not powered to detect small effects; findings will be used to estimate effect sizes and assess feasibility for a future larger-scale trial.

DETAILED DESCRIPTION:
This study investigates whether incorporating an indirect contact component into an existing school-based mental health literacy (MHL) program enhances reductions in stigma-specifically vignette-based social distance-among elementary school students. Indirect contact is implemented through a teacher-delivered story describing the lived experience and recovery of a well-known soccer player who publicly disclosed his mental illness. This approach aims to promote empathy, reduce negative stereotypes, and strengthen intentions to seek or recommend appropriate help.

The study uses a cluster-randomized parallel-group design, with four 5th-grade classes assigned (2:2) to either the intervention or control condition. Both groups receive a standardized 45-minute MHL lesson including an animated educational video and discussion materials. The intervention arm additionally receives the indirect contact component within the same 45-minute period. The lesson is delivered by classroom teachers.

Assessments occur at three time points:

* T1 (baseline): before the lesson
* T2 (post-test): immediately after the lesson
* T3 (follow-up): 2-3 months after the lesson

The primary outcome is a 5-item social distance scale based on a vignette ("A-san") describing symptoms consistent with depression. Secondary outcomes include:

* mental health knowledge
* intentions to support a friend with similar problems
* perceived need for help
* personal help-seeking intentions
* intended help-seeking sources

Because this is a pilot trial, the goals are to evaluate feasibility (recruitment, retention, acceptability, implementation fidelity) and to estimate preliminary effect sizes to inform sample size calculations for a future fully powered cluster randomized trial. After T3 data collection, students in the control arm will be offered an educational supplement that includes the indirect contact story.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in 5th grade at one of the eight participating public elementary schools in Kanazawa, Japan.
* Aged 10-11 years old.
* Passive consent obtained from guardians; verbal assent obtained from children.
* Able to complete self-report questionnaires.

Exclusion Criteria:

* Students whose parents/guardians opted out of the study.

Note: Students who were absent on the day of the pre-test (T1) were excluded from the analysis population but not from the initial study cohort.

Ages: 10 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Social Distance Scale Score (Stigma) | Baseline (T1), immediately post-intervention (T2), and 3-month follow-up (T3)
  A 5-item scale adapted from the Social Distance Scale using a vignette format. Each item rated on a 4-point scale (1=definitely willing to 4=definitely unwilling), total score range 4-20. Higher scores indicate greater stigma. Cronbach's alpha was 0.88.

SECONDARY OUTCOMES:
Mental Health Knowledge Score | Baseline (T1), immediately post-intervention (T2), and 3-month follow-up (T3)
  An 8-item true/false questionnaire developed based on the SMHLP content. Scores range from 0 to 8, with higher scores indicating greater knowledge about mental health and illnesses. Cronbach's alpha was 0.65.
Help-Seeking Intention | Baseline (T1), immediately post-intervention (T2), and 3-month follow-up (T3)
  A vignette-based item asking whether students themselves would seek help if they were experiencing similar mental health difficulties. Responses were on a 4-point scale: "Definitely yes", "Probably yes", "Probably not", and "Definitely not". Students were considered to have the intention to seek help if they responded "Definitely yes".
Recognition of the necessity to seek help | Baseline (T1), immediately post-intervention (T2), and 3-month follow-up (T3)
  A single vignette-based item asking whether students thought the character in the scenario should seek help from others. Responses were on a 4-point scale: "Definitely yes", "Probably yes", "Probably not", and "Definitely not". Students were considered to recognize the necessity to seek help when they responded "Definitely yes".
Intention to Help Peers | Baseline (T1), immediately post-intervention (T2), and 3-month follow-up (T3)
  Students were asked to rate their likelihood of performing various desirable supportive behaviors for a peer in distress. Each item was rated on a 4-point scale. Students were considered to have the intention to help if they selected "Definitely yes" for at least one of the behaviors. An example of a behavior is: "I would ask about or listen to their story to understand their situation in detail."

IPD SHARING:
Plan to Share IPD: No
Because this study involves minors in a school-based setting and includes sensitive educational and mental health-related information, individual participant data cannot be shared. Disclosure of such data could risk re-identification even after de-identification procedures. In accordance with ethical guidelines and institutional policies, IPD will not be made available.